CLINICAL TRIAL: NCT01445522
Title: A Phase I Study of ABT-888 in Combination With Metronomic Cyclophosphamide in Adults With Refractory Solid Tumors and Lymphomas
Brief Title: ABT-888 Plus Metronomic Cyclophosphamide to Treat Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 090048; 09-C-0048; NCT00810966 (obsolete NCT alias)
Record Dates: First submitted 2011-09-30; First posted 2011-10-03 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2012-06-29

CONDITIONS: Neoplasms; Lymphoma
Keywords: PARP Inhibitor; DNA Damage; Chemotherapy; Advanced Cancer; DNA Repair
MeSH Terms: conditions — Neoplasms; Lymphoma | interventions — veliparib; Cyclophosphamide

INTERVENTIONS:
Drug: ABT-888
Drug: Cyclophosphamide

SUMMARY:
Background:

* Cyclophosphamide (CP) is a drug approved by the Food and Drug Administration for the treatment of certain cancers. It works by causing DNA damage, resulting in cell death, including cancer cells.
* ABT-888 is an experimental drug that has been given to a small number of patients. It works by preventing DNA repair in tumor cells.

Objectives:

* To test the safety of the combination of ABT-888 and CP, and to determine the dose of each drug that can be given together to patients with cancer.
* To see how the body handles ABT-888 when given together with CP
* To evaluate the anti-tumor response of the drug combination.

Eligibility:

* Adults with solid tumors or lymphoid cancers (lymphoma and chronic lymphocytic leukemia) whose disease does not respond to standard treatments.

Design:

* Patients take ABT-888 by mouth once a day for 7, 14 or 21 days, depending on the dose level assigned to the individual patient.
* Patients take CP by mouth once a day every day in 21-day cycles. (Some patients take CP for 14 days only.)
* Patients undergo tests and procedures periodically during the study, including:
* Clinic visit and physical examination at the beginning of each cycle
* Blood and urine tests, electrocardiogram, measurement of vital signs
* CT scans, MRI scans or ultrasound tests to check the response of the tumor to treatment
* Tumor biopsies (optional)
* Bone marrow aspiration and biopsy

DETAILED DESCRIPTION:
Background:

* The poly (ADP-ribose) polymerase (PARP) family of enzymes is characterized by the ability to poly-ADP-ribosylate protein substrates. PARP-1 and PARP-2 play a critical role in the maintenance of genomic stability by regulating a variety of DNA repair mechanisms.
* PARP activity has been shown to be important in base excision repair pathways. The inhibition of PARP could inhibit the repair of the DNA damage caused by alkylating agents such as cyclophosphamide. ABT-888 has been shown to potentiate the action of cyclophosphamide in xenografts models. ABT-888 is an orally delivered PARP inhibitor and cyclophosphamide can be delivered orally as an alkylating agent.
* Metronomic therapy with cyclophosphamide has demonstrated efficacy in multiple tumor types including, but not limited to, ovarian cancer, lymphoma, prostate cancer, and breast cancer. Its activity has been at least partially attributed to mediation of anti-angiogenic effects through induction of apoptosis in endothelial cells.

Objectives:

* Establish the safety and tolerability of the combination of ABT-888 with metronomic cyclophosphamide in patients with refractory solid tumors and lymphomas.
* Establish the maximum tolerated dose (MTD) of the combination of ABT-888 with metronomic cyclophosphamide.
* Evaluate the pharmacokinetics of ABT-888 when administered combination with cyclophosphamide.
* Evaluate for anti-tumor response.
* Determine the effects of the study treatment on the level of PARP inhibition and gamma-H2AX in PBMCs and tumor samples.

Eligibility:

* Patients with histologically documented solid tumors or lymphoid malignancies (lymphoma and CLL) whose disease has progressed following standard therapy or who have no acceptable standard treatment options.
* No major surgery, radiation or chemotherapy within four weeks prior to study enrollment, and recovered from toxicities of prior therapies to at least eligibility levels.

Study Design:

* ABT-888 will be administered orally once daily for 7 to 21 days, depending on the dose level (see below). Cyclophosphamide will be administered orally once daily in 50 mg or 100 mg doses continuously from days 1 to 21. Cycle length is 21 days.
* Dose escalation will proceed as outlined below. Once MTD is established, 6 additional patients will be enrolled at the MTD to evaluate that dose further and extend PD studies at that dose level.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Patients with histologically documented solid tumors or lymphoid malignancies (lymphoma and CLL) refractory to standard therapy or who have no acceptable standard treatment options. Patients with lymphoid malignancies will be eligible if their disease has progressed following standard therapy and if stem cell transplantation is not indicated or has been refused.
* Any prior therapy must have been completed greater than or equal to 4 weeks (greater than 6 weeks for nitrosoureas or mitomycin C) prior to enrollment on protocol, and the participant must have recovered to eligibility levels (CTCAE Grade less than or equal to 1) from prior toxicity. Prior radiation should have been completed greater than or equal to 4 weeks prior to study enrollment, and all associated toxicities should have resolved to eligibility levels. Patients must be greater than or equal to 2 weeks since any investigational agent administered as part of a Phase 0 study, and should have recovered to eligibility levels from any toxicities.
* Age greater than or equal to 18 years. Because no dosing or adverse event data are currently available on the use of ABT-888 in patients less than 18 years of age, children are excluded from this study, but may be eligible for future pediatric Phase I combination trials.
* Karnofsky performance status greater than or equal to 60%, see Appendix A.
* Life expectancy of greater than 3 months.
* Patients must have normal organ and marrow function as defined below:

  * absolute neutrophil count greater than or equal to 1,500/microL (mcL)
  * platelets greater than or equal to 100,000/microL (mcL)
  * total bilirubin less than 1.5 times the institutional upper limit of normal
  * AST(SGOT)/ALT(SGPT) less than or equal to 2.5 times the institutional upper limit of normal
  * creatinine less than 1.5 times the institutional upper limit of normal

OR

creatinine clearance greater than or equal to 60 mL/min for patients with creatinine levels 1.5 times the institutional upper limit of normal.

* The effects of ABT-888 on the developing human fetus are unknown. For this reason and because cyclophosphamide hydrochloride used in this trial is known to be teratogenic, women of childbearing potential and men must agree to use adequate contraception (abstinence; female use of hormonal methods, or barrier methods of birth control; male use of a condom) prior to study entry, for the duration of study participation, and for 3 months after completion of study. Because there is a risk for adverse events in nursing infants secondary to treatment of the mother with cyclophosphamide, breastfeeding should be discontinued while the patient is on this trial and for 30 days after completion of treatment on this trial. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Ability to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

- Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier. Patients must be greater than or equal to 2 weeks since any investigational agent administered as part of a Phase 0 study, and should have recovered to eligibility levels from any toxicities.

Patients who have been administered ABT-888 as part of a single or limited dosing study, such as a Phase 0 study, should not be excluded from participating in this study solely because of receiving prior ABT-888.

Patients who have received prior cyclophosphamide should not be excluded solely because of receiving prior cyclophosphamide.

* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Patients with gliomas, symptomatic CNS metastases or carcinomatous meningitis are excluded from this clinical trial. Patients with history of CNS metastases who have received treatment and whose CNS metastatic disease status has remained stable for greater than or equal to 3 months without steroids or anti-seizure medications may be eligible. These patients may be enrolled at the discretion of the principal investigator.
* Patients with a history of seizures.
* Patients with HIV who are taking protease inhibitors.
* Patients with gastrointestinal conditions that might predispose for drug intolerability or poor drug absorption (e.g., inability to take oral medication or a requirement for IV alimentation, prior surgical procedures affecting absorption, malabsorption syndrome, active peptic ulcer disease) are excluded. Subjects with ulcerative colitis, inflammatory bowel disease, or a partial or complete small bowel obstruction are also excluded.

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2008-12-03; Primary Completion 2012-07-03 (Actual); Study Completion 2012-07-03 (Actual)

PRIMARY OUTCOMES:
Establish the safety and tolerability of the combination of ABT-888 with metronomic cyclophosphamide in patients with refractory solid tumors and lymphomas. Establish the MTD of the combination of ABT-888 with metronomic cyclophosphamide.

SECONDARY OUTCOMES:
Evaluate the pharmacokinetics of ABT-888 when administered combination with cyclophosphamide. Evaluate for anti-tumor response.

CONTACTS AND LOCATIONS:
Overall Officials: Shivaani Kummar, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (2):
- United States (2):
  - City of Hope National Medical Center, Duarte, California
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland

REFERENCES:
- [Background] Alderson T. New targets for cancer chemotherapy--poly(ADP-ribosylation) processing and polyisoprene metabolism. Biol Rev Camb Philos Soc. 1990 Nov;65(4):623-41. doi: 10.1111/j.1469-185x.1990.tb01240.x. No abstract available. PMID 2124932
- [Background] Ame JC, Rolli V, Schreiber V, Niedergang C, Apiou F, Decker P, Muller S, Hoger T, Menissier-de Murcia J, de Murcia G. PARP-2, A novel mammalian DNA damage-dependent poly(ADP-ribose) polymerase. J Biol Chem. 1999 Jun 18;274(25):17860-8. doi: 10.1074/jbc.274.25.17860. PMID 10364231
- [Background] Ame JC, Spenlehauer C, de Murcia G. The PARP superfamily. Bioessays. 2004 Aug;26(8):882-93. doi: 10.1002/bies.20085. PMID 15273990